CLINICAL TRIAL: NCT01473537
Title: A Double Blind, Randomized, Cross Over Designed Trial of Fluoride Prevention by Double Rinse With Calcium and Fluoride
Brief Title: Optimised Fluoride Prevention by Double Rinse With Fluoride and Calcium
Acronym: Fluor-Ca
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gunilla Sandborgh Englund, professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DDM 2011/1; 2011-001885-16 (EudraCT Number)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Dental Caries
Keywords: dental caries/prevention and control; oral health; cariostatic agents
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- calcium lactate solution 75 mM (Active Comparator)
  Interventions: Drug: calcium lactate solution
- calcium lactate solution 150 mM (Active Comparator)
  Interventions: Drug: calcium lactate solution
- placebo (Placebo Comparator)
  Interventions: Drug: calcium lactate solution

INTERVENTIONS:
Drug: calcium lactate solution — Calcium lactate solution 75 mM, 150 mM, 175 mM and placebo

SUMMARY:
Aim: to determine the optimal Ca2+ concentration with 905 ppm F as NaF. Study design: Experimental study in 10 volunteers. Single blind mouth rinse with calcium lactate solution (150; 75; 0 mM Ca-lactate) is immediately followed by a standard fluoride rinse.

Procedure: Rinses are performed in the evening. The rinse combinations are given in a random order, and the subjects are unaware of the sequence. At least 3 days separates the use of each rinse. Dosage: 20 mL and 1 minute rinse with each solution.

Saliva samples: Twelve hours after rinsing, unstimulated saliva samples are collected by expectoration.

Analysis: The fluoride concentration in saliva samples are analysed Statistics and data handling: Fluoride in saliva 12 hours after rinsing are examined by one-way ANOVA, repeated measures design.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* 10 natural teeth or more
* willing to refrain from use of fluoride containing products
* signed informed consent

Exclusion Criteria:

* less than 10 natural teeth
* reduced cognitive skills
* does not speak and/or understand Swedish
* ongoing oral or systemic infections
* pregnancy
* breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fluoride concentration in resting saliva | 12 hours after rinse

SECONDARY OUTCOMES:
Discomfort by calcium lactate rinse | 12 hours after rinse

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Sandborgh-Englund, Prof, DDS, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Dept Dental Medicine, Huddinge, Sweden